CLINICAL TRIAL: NCT00838097
Title: A Prospective Registry Study Observing the Safety and Patterns of Use of Darbepoetin Alfa in EU Paediatric Chronic Kidney Disease Patients Receiving or Not Receiving Dialysis
Brief Title: European Union Registry in Paediatric Chronic Kidney Disease Patients Looking at Safety and Usage Patterns of Darbepoetin Alfa
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20070211
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease
Keywords: CKD; Paediatric; Darbepoetin Alfa
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (1):
- Darbepoetin alfa: Participants with chronic kidney disease who received darbepoetin alfa for the treatment of anaemia as part of routine clinical practice.

SUMMARY:
This European study observes paediatric patients with Chronic Kidney Disease using Darbepoetin Alfa to assess the drug's long term safety and profile the patterns of its use within this population.

ELIGIBILITY:
Inclusion Criteria:

* Anaemia attributed to Chronic Kidney Disease (CKD)
* Sixteen years of age or under
* Documented CKD as demonstrated by estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m² (Schwartz equation) for ≥3 months if not on dialysis, or: Receiving dialysis
* Treatment with darbepoetin alfa
* Documented informed consent by a parent or authorised individual, if required, and assent by the patient if appropriate

Exclusion Criteria:

* Active malignancy or current chemotherapy or radiation therapy
* Investigator unlikely to be able to obtain adequate follow-up information, or participant will not be available for follow-up assessment
* Currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study; subject receiving other investigational agents

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Specialist Centres
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on 26 February 2008; last participant was enrolled on 24 February 2011.
Period: Overall Study
Arm/Group | Darbepoetin Alfa
Started | 321
Received Darbepoetin Alfa | 319
Completed | 145
Not Completed | 176
Not completed — Ineligibility determined | 6
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 3
Not completed — Requirement for alternative therapy | 2
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 11
Not completed — Death | 6
Not completed — Protocol-specified criteria | 142

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who received at least 1 dose of darbepoetin alfa during the study.
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (5.0)
Age, Customized [Number; unit: participants]
  < 1 year | 13
  1 to < 6 years | 83
  6 to < 12 years | 90
  ≥ 12 years | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 177
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 274
  Black or African American | 9
  Asian | 8
  Japanese | 0
  Other | 9
  Not recorded | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Drug Reactions (SADR), Serious Adverse Events (SAEs) or Events of Medical Interest (EMIs)
Description: An ADR was defined as an undesirable medical occurrence or worsening of a pre-existing medical condition that the investigator considered associated with the use of darbepoetin alfa. An AE is any untoward medical occurrence or worsening of a pre-existing condition whether or not considered to have a causal relationship with darbepoetin alfa. An SADR or SAE is any ADR or AE that is either: • Fatal • Life threatening • Requires or prolongs in-patient hospitalization • A persistent or significant disability/incapacity, or • A congenital anomaly/birth defect. An EMI is defined as one of the following pre-specified AEs: Thromboembolic Events (eg, venous thrombosis, embolism, vascular occlusion) • Seizures • Severe hypertension (Investigator discretion accompanied by recorded blood pressure) • Cardiovascular events (eg, cardiac arrhythmia, myocardial ischaemia/infarction, heart failure) • Pure red cell aplasia (PRCA) • Hypersensitivity reactions (eg, rash, urticaria, anaphylaxis).
Time Frame: 2 years
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 319
participants
  Serious Adverse Drug Reactions | 4
  Serious Adverse Events | 162
  Events of Medical Interest | 39

2. Secondary Outcome: Hemoglobin Concentration by Three Monthly Intervals
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 319
g/dL
  Baseline (n=308) | 11.06 (1.62) [10.88 to 11.24]
  Month 3 (n=260) | 11.47 (1.64) [11.27 to 11.67]
  Month 6 (n=269) | 11.34 (1.32) [11.18 to 11.50]
  Month 9 (n=245) | 11.43 (1.50) [11.24 to 11.62]
  Month 12 (n=214) | 11.39 (1.38) [11.21 to 11.58]
  Month 15 (n=199) | 11.26 (1.35) [11.08 to 11.45]
  Month 18 (n=167) | 11.30 (1.50) [11.08 to 11.53]
  Month 21 (n=154) | 11.30 (1.34) [11.09 to 11.51]
  Month 24 (n=151) | 11.42 (1.40) [11.20 to 11.65]

3. Secondary Outcome: Weight Adjusted Darbepoetin Alfa Monthly Dose by Monthly Intervals
Description: Baseline dose = the daily dose equivalent x 30, where the daily dose equivalent = the last available dose prior to or at Day 1 / reported intended frequency.
Time Frame: Baseline and Months 1 to 24
Population: Full analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: μg/kg/month
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 319
μg/kg/month
  Baseline (n=273) | 1.99 [1.82 to 2.18]
  Month 1 (n=311) | 1.90 [1.74 to 2.07]
  Month 2 (n=304) | 1.91 [1.75 to 2.09]
  Month 3 (n=297) | 1.94 [1.76 to 2.14]
  Month 4 (n=287) | 1.87 [1.69 to 2.07]
  Month 5 (n=277) | 1.82 [1.65 to 2.02]
  Month 6 (n=269) | 1.87 [1.69 to 2.08]
  Month 7 (n=256) | 1.79 [1.60 to 2.00]
  Month 8 (n=245) | 1.79 [1.61 to 1.98]
  Month 9 (n=233) | 1.69 [1.52 to 1.89]
  Month 10 (n=227) | 1.63 [1.47 to 1.82]
  Month 11 (n=216) | 1.72 [1.53 to 1.92]
  Month 12 (n=211) | 1.66 [1.49 to 1.85]
  Month 13 (n=206) | 1.58 [1.40 to 1.78]
  Month 14 (n=200) | 1.65 [1.46 to 1.86]
  Month 15 (n=193) | 1.71 [1.52 to 1.94]
  Month 16 (n=186) | 1.71 [1.51 to 1.93]
  Month 17 (n=180) | 1.73 [1.54 to 1.96]
  Month 18 (n=170) | 1.71 [1.51 to 1.94]
  Month 19 (n=164) | 1.71 [1.50 to 1.95]
  Month 20 (n=162) | 1.70 [1.48 to 1.96]
  Month 21 (n=157) | 1.79 [1.56 to 2.05]
  Month 22 (n=155) | 1.70 [1.46 to 1.97]
  Month 23 (n=154) | 1.63 [1.41 to 1.88]
  Month 24 (n=146) | 1.44 [1.22 to 1.69]

4. Secondary Outcome: Parathyroid Hormone Level by Three Monthly Intervals
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 319
pmol/L
  Baseline (n=228) | 20.44 (1.62) [11.82 to 36.81]
  Month 3 (n=236) | 19.76 (1.64) [9.93 to 36.70]
  Month 6 (n=246) | 18.12 (1.32) [9.87 to 29.40]
  Month 9 (n=225) | 16.70 (1.50) [9.20 to 33.60]
  Month 12 (n=194) | 19.11 (1.38) [8.55 to 33.50]
  Month 15 (n=184) | 17.51 (1.35) [9.57 to 30.67]
  Month 18 (n=150) | 17.69 (1.50) [9.56 to 36.23]
  Month 21 (n=142) | 18.12 (1.34) [8.93 to 36.75]
  Month 24 (n=137) | 21.20 (1.40) [11.13 to 35.79]

5. Secondary Outcome: Number of Participants With Non-serious Adverse Drug Reactions (ADRs)
Description: An ADR was defined as an undesirable medical occurrence or worsening of a pre-existing medical condition that the investigator considered associated with the use of darbepoetin alfa. A non-serious ADR was one in which none of the following applied:
  * Fatal
  * Life threatening
  * Required or prolonged in-patient hospitalization
  * A persistent or significant disability/incapacity, or
  * A congenital anomaly/birth defect.
Time Frame: 2 years
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 319
participants | 4

ADVERSE EVENTS:
Time Frame: 2 years
Description: In this study only adverse drug reactions, serious adverse events and events of medical interest were collected. Other Adverse Events summarizes the non-serious occurrences of adverse drug reactions and non-serious occurrences of events of medical interest that exceed the indicated frequency threshold.
Arm/Group | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 162/319
Other Adverse Events (participants affected / at risk) | 7/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=319)
Anaemia (Blood and lymphatic system disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Congenital mitochondrial cytopathy (Congenital, familial and genetic disorders) | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 1
Autoimmune thyroiditis (Endocrine disorders) | 1
Goitre (Endocrine disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Blindness (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Catheter site haematoma (General disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Device malfunction (General disorders) | 1
Hyperthermia (General disorders) | 1
Medical device complication (General disorders) | 4
Oedema (General disorders) | 1
Pyrexia (General disorders) | 4
Thrombosis in device (General disorders) | 2
Acute hepatic failure (Hepatobiliary disorders) | 1
Kidney transplant rejection (Immune system disorders) | 2
Arteriovenous fistula site infection (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 6
Bronchitis viral (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 6
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 6
Device related sepsis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Fungal peritonitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 19
Gastroenteritis norovirus (Infections and infestations) | 2
Gastroenteritis rotavirus (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Keratitis herpetic (Infections and infestations) | 1
Leishmaniasis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 32
Peritonitis bacterial (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 6
Pseudomonal sepsis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 6
Pyelonephritis acute (Infections and infestations) | 4
Respiratory tract infection (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 7
Urosepsis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral infection (Infections and infestations) | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 5
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Transplant failure (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 4
Blood urea increased (Investigations) | 1
Cardiac output increased (Investigations) | 1
HLA marker study positive (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Fluid overload (Metabolism and nutrition disorders) | 3
Fluid retention (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypervolaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 10
Epilepsy (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Migraine with aura (Nervous system disorders) | 1
Neuritis (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Anuria (Renal and urinary disorders) | 1
Bladder dysfunction (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 7
Renal impairment (Renal and urinary disorders) | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 2
Urinary tract disorder (Renal and urinary disorders) | 1
Vesicoureteric reflux (Renal and urinary disorders) | 1
Priapism (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Inadequate diet (Social circumstances) | 1
Accelerated hypertension (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 13
Hypertensive crisis (Vascular disorders) | 5
Hypertensive emergency (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Thrombophlebitis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=319)
Injection site pain (General disorders) | 4
Drug hypersensitivity (Immune system disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.